CLINICAL TRIAL: NCT05354986
Title: Impact of a Newly Formulated Tooth Paste in the Prevention/Elimination of Tooth Staining Associated With Adjunctive Use Chlorhexidine Mouth Rinses to Subgingival Instrumentation. A Randomized Clinical Trial
Brief Title: Impact of a Newly Formulated Toothpaste in Tooth Staining Associated With Chlorhexidine Rinses
Acronym: PaSTaining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Dentaid SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 68-071021; 21/546-EC_X (Other: Comité Ético Hospital Clínico San Carlos)
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-07

CONDITIONS: Tooth Staining; Periodontitis
Keywords: Tooth staining; Periodontitis; Chlorhexidine; tripolyphosphate and polyvinylpyrrolidone (PVP)
MeSH Terms: conditions — Tooth Discoloration; Periodontitis | interventions — Toothpastes; hexametaphosphate; triphosphoric acid; Povidone

STUDY DESIGN:
Intervention Model Description: Two consecutive parallel, double-blind, randomized, placebo-controlled, 2-week, clinical trials
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: test and placebo toothpastes would be identical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control-Control (Placebo Comparator): Immediately after the second session of subgingival instrumentation (initial visit, RCT #1) subjects will be randomly assigned to one of two groups, test or placebo.
  0-2 weeks: The control group will use three times daily a provided manual toothbrush with the placebo toothpaste (identical to the test tooth paste, but without the active ingredients), followed by the use, twice daily, of a 0.12% chlorhexidine mouth rinse.
  Subjects will stop using the mouth rinse, and will start the second RCT, being randomized again, within each group of the first RCT, to the placebo or test toothpaste.
  2-4 weeks: The control group will use three times daily a provided manual toothbrush with the placebo toothpaste (identical to the test tooth paste, but without the active ingredients), followed by the use, twice daily, of a 0.12% chlorhexidine mouth rinse.
  Interventions: Other: Toothpaste without hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP)
- Control-test (Experimental): Immediately after the second session of subgingival instrumentation (initial visit, RCT #1) subjects will be randomly assigned to one of two groups, test or placebo.
  0-2 weeks: The control group will use three times daily a provided manual toothbrush with the placebo toothpaste (identical to the test tooth paste, but without the active ingredients), followed by the use, twice daily, of a 0.12% chlorhexidine mouth rinse.
  Subjects will stop using the mouth rinse, and will start the second RCT, being randomized again, within each group of the first RCT, to the placebo or test toothpaste.
  2-4 weeks: The experimental group will use three times daily a provided manual toothbrush with the test toothpaste (Dentaid, Barcelona, Spain), followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Interventions: Other: Toothpaste with hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP)
- Test-control (Experimental): Immediately after the second session of subgingival instrumentation (initial visit, RCT #1) subjects will be randomly assigned to one of two groups, test or placebo.
  0-2 weeks: The experimental group will use three times daily a provided manual toothbrush with the test toothpaste (Dentaid, Barcelona, Spain), followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Subjects will stop using the mouth rinse, and will start the second RCT, being randomized again, within each group of the first RCT, to the placebo or test toothpaste.
  2-4 weeks: The control group will use three times daily a provided manual toothbrush with the placebo toothpaste (identical to the test tooth paste, but without the active ingredients), followed by the use, twice daily, of a 0.12% chlorhexidine mouth rinse.
  Interventions: Other: Toothpaste with hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP)
- Test-test (Experimental): Immediately after the second session of subgingival instrumentation (initial visit, RCT #1) subjects will be randomly assigned to one of two groups, test or placebo.
  0-2 weeks: The experimental group will use three times daily a provided manual toothbrush with the test toothpaste (Dentaid, Barcelona, Spain), followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Subjects will stop using the mouth rinse, and will start the second RCT, being randomized again, within each group of the first RCT, to the placebo or test toothpaste.
  2-4 weeks: The experimental group will use three times daily a provided manual toothbrush with the test toothpaste (Dentaid, Barcelona, Spain), followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Interventions: Other: Toothpaste with hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP)

INTERVENTIONS:
Other: Toothpaste with hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP) — Subgingival instrumentation will be performed in two sessions, with a maximum interval of one week, with hand and automatic devices, under local anaesthesia. Full-mouth dental polishing (air-polishing) will be performed immediately after the second session, to eliminate any dental staining.
  Experimental anti-staining toothpaste formulation (Dentaid, Barcelona, Spain) includes hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP), within its ingredients. Participants will use the test or control toothpaste three times daily with a manual toothbrush followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Arms: Control-test; Test-control; Test-test
Other: Toothpaste without hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP) — Subgingival instrumentation will be performed in two sessions, with a maximum interval of one week, with hand and automatic devices, under local anaesthesia. Full-mouth dental polishing (air-polishing) will be performed immediately after the second session, to eliminate any dental staining.
  Experimental anti-staining toothpaste formulation without tripolyphosphate and polyvinylpyrrolidone (PVP), within its ingredients. Participants will use the test or control toothpaste three times daily with a manual toothbrush followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
  Arms: Control-Control

SUMMARY:
Dental staining may interfere with compliance with chlorhexidine mouth rinse use

Thus, developing strategies to control tooth staining associated with chlorhexidine use may be relevant for improving compliance. Thus, a new anti-staining toothpaste formulation (Dentaid, Barcelona, Spain) has been recently developed, aiming to interfere with the development of extrinsic staining associated with chlorhexidine use (preventive action), but also with the capacity of removing staining already formed. For that, the proposed formulation includes hexametaphosphate, tripolyphosphate and polyvinylpyrrolidone (PVP), within its ingredients. Thus, it may be relevant to test the efficacy of this new anti-staining toothpaste formulation in two consecutive randomized clinical trials (RCTs).

Objectives The primary objective of these RCTs will be to evaluate the capacity of preventing tooth staining, associated with the use of a chlorhexidine mouth rinse, adjunctive to subgingival instrumentation (step 2 of periodontal therapy) (RCT #1). As secondary objective, the capacity of eliminating or reducing tooth staining already present will be assessed (RCT #2).

DETAILED DESCRIPTION:
The primary objective of these RCTs will be to evaluate the capacity of preventing tooth staining, associated with the use of a chlorhexidine mouth rinse, adjunctive to subgingival instrumentation (step 2 of periodontal therapy) (RCT #1). As secondary objective, the capacity of eliminating or reducing tooth staining already present will be assessed (RCT #2).

Additional objectives will include to test: (1) the safety of the tested formulation, in terms of adverse events and tolerability; (2) patient´s evaluation of the product, by means of patient-reported outcome measures (PROMs); and (3) clinical impact of the tested formulation in terms of periodontal clinical outcomes.

Consecutive subjects, referred to the Post-Graduate Periodontal Clinic in the University Complutense, Madrid, seeking for treatment of periodontitis in stages I-III will be screened, and enrolled in the clinical trials if they fulfil the following criteria and accept to participate by filling an informed consent

Two consecutive parallel, double-blind, randomized, placebo-controlled, 2-week, clinical trials have been designed.

Screening visit After completing a questionnaire including the subject's medical health status, medication and smoking habit [smoker defined when currently smoking ≥ 9 cigarettes per day], a careful oral health evaluation will be carried out. If subjects met the inclusion/exclusion criteria, the investigator will inform them about the aims and details of the study and will request their voluntary participation. Once they accept, by signing the Institutional Review Board (IRB) approved informed consent form, they will be enrolled in the study.

Pre-treatment visit At this visit the oral health of each participant, identified by a unique trial number, will be examined. Clinical parameters will be recorded around all teeth, except the third molars.

Treatment visits All interventions, included in the steps 1 and 2 of periodontal therapy will be implemented according to the patient´s needs. Specifically, subgingival instrumentation will be performed in two sessions, with a maximum interval of one week, with hand and automatic devices, under local anaesthesia. Full-mouth dental polishing (air-polishing) will be performed immediately after the second session, to eliminate any dental staining.

Immediately after the second session of subgingival instrumentation (initial visit, RCT #1) subjects will be randomly assigned to one of two groups, test or placebo. Randomization will be performed using true random numbers from a computer-generated list, stratified for tobacco smoking (smokers of 10 or more cigarettes per day versus other smokers, former smokers and non-smokers):

1. The experimental group will use three times daily a provided manual toothbrush with the test toothpaste (Dentaid, Barcelona, Spain), followed by the use, twice daily, of a 0.12% chlorhexidine, commercially available, mouth rinse.
2. The control group will use three times daily a provided manual toothbrush with the placebo toothpaste (identical to the test tooth paste, but without the active ingredients), followed by the use, twice daily, of a 0.12% chlorhexidine mouth rinse,

All subjects will be masked to their group allocation and will receive their assigned products kit containing: a manual toothbrush (Vitis Suave, Dentaid, Barcelona, Spain), the test or placebo toothpaste, and the mouth rinse with dose caps. They will be instructed to brush with the toothpaste (the amount of a pee size) for 2 minutes, twice daily, and then rinse for 30 seconds with 15 mL of the mouth rinse, twice daily. Standardized instructions will be given for mechanical supragingival biofilm control, including the use of interdental brushes (Interprox®, Dentaid, Barcelona, Spain). Each subject will receive standardized verbal and written instructions on how to use the assigned products.

2-week visit (final visit, RCT #1; initial visit, RCT #2) Two weeks after the second session of subgingival instrumentation, an oral examination will be performed to evaluate possible adverse effect, and dental plaque index will be recorded. Clinical photographs will be also taken to assess staining (four, for sextants 2 and 5, for buccal and palatal surfaces).

The subjects will be asked about the occurrence of any adverse effects. A questionnaire on product usage and perceptions (PROMs), dietary habits and compliance with product use will be filled by the patients. The study coordinator will collect the empty and unused tubes and bottles. Subjects will be provided with a new kit containing the necessary assigned products.

Subjects will stop using the mouth rinse, and will start the second RCT, being randomized again, within each group of the first RCT, to the placebo or test toothpaste. Thus, at the 2-week visit, half of each group will continue with the same toothpaste and the other half will change toothpaste, creating four different groups, when considering both RCTs: group control-control, group control-test, group test-control, group test-test)

4-week visit (final visit, RCT #2) After 4 weeks, a comprehensive oral examination will be performed, including the assessment of clinical variables. The subjects will be asked about the occurrence of any adverse effects and the study coordinator will collect the empty and unused tubes. A new questionnaire on product usage and perceptions (PROMs), dietary habits and compliance with product use will be filled by the patients.

Clinical photographs (four, for sextants 2 and 5, for buccal and palatal surfaces) will be also taken to assess staining. All subjects will be provided with a professional dental prophylaxis at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 30-69 years old.
* Periodontitis patients, in stages I-III, requiring steps 1 and 2 of periodontal treatment including full-mouth subgingival instrumentation.
* Systemically healthy, following the criteria of the American Society of Anesthesiologists (ASA), for patients ASA type I or II (see also exclusion criteria).
* Presence of at least three evaluable teeth in each quadrant.
* No orthodontic banding or removable prosthesis.
* Subjects willing to participate and comply with the requirements of the study.

Exclusion Criteria:

* Acute periodontal conditions.
* Antibiotic intake within the previous month.
* Chronic use of analgesic or anti-inflammatory drugs.
* Pregnant women.
* Any adverse medical history (diabetes, osteoporosis, immunosuppression…) or long-term medication (chemotherapy and immunosuppression treatment; pharmacological treatment associated with gingival overgrowth such as the use of phenytoin, phenobarbital, lamotrigine, vigabatrin, ethosuximide, topiramate, primidone, nifedipine, amlodipine, verapamil, cyclosporine) influencing gingival conditions.
* Conditions which require antibiotic prophylaxis (infectious endocarditis, cardiac valve prosthesis…).

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Tooth Staining | 2 weeks
  GRÜNDEMANN MODIFIED STAIN INDEX (GMSI) (Gründemann et al., 2000). 2. Photographs of buccal and lingual/palatal areas of lower and upper anterior teeth, from canine to canine.
  The zones to be scored, buccal only:
  Mesial (A), Distal (A), Gingival (G) and Incisal (I)
  The intensity in each zone will be scored using the following criteria described by Lobene (Lobene, 1968):
  Score=0 No stain Score=1 Light stain Score=2 Moderate stain Score=3 Heavy stain
Tooth Staining | 4 weeks
  GRÜNDEMANN MODIFIED STAIN INDEX (GMSI) (Gründemann et al., 2000). 2. Photographs of buccal and lingual/palatal areas of lower and upper anterior teeth, from canine to canine.
  The zones to be scored, buccal only:
  Mesial (A), Distal (A), Gingival (G) and Incisal (I)
  The intensity in each zone will be scored using the following criteria described by Lobene (Lobene, 1968):
  Score=0 No stain Score=1 Light stain Score=2 Moderate stain Score=3 Heavy stain

SECONDARY OUTCOMES:
Dental plaque | 0 weeks
  Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962). Scale: 0-5.
  Score=0 No Plaque Score=1 The presence of a discontinuous line of plaque at the gingival margin e.g. small islands Score=2 A continuous line of plaque at the gingival margin which does not extend greater than 1 mm from the margin Score=3 Plaque coverage which is greater than 1 mm but does not extend more than one third of the tooth Score=4 Plaque which covers more than one third but not more than two third of the tooth surface Score=5 Plaque coverage over more than two third of the tooth surface.
Dental plaque | 2 weeks
  Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962) Score=0 No Plaque Score=1 The presence of a discontinuous line of plaque at the gingival margin e.g. small islands Score=2 A continuous line of plaque at the gingival margin which does not extend greater than 1 mm from the margin Score=3 Plaque coverage which is greater than 1 mm but does not extend more than one third of the tooth Score=4 Plaque which covers more than one third but not more than two third of the tooth surface Score=5 Plaque coverage over more than two third of the tooth surface.
Dental plaque | 4 weeks
  Turesky et al. (Turesky, Gilmore, & Glickman, 1970) modification of the Quigley and Hein index (Quigley & Hein, 1962) Score=0 No Plaque Score=1 The presence of a discontinuous line of plaque at the gingival margin e.g. small islands Score=2 A continuous line of plaque at the gingival margin which does not extend greater than 1 mm from the margin Score=3 Plaque coverage which is greater than 1 mm but does not extend more than one third of the tooth Score=4 Plaque which covers more than one third but not more than two third of the tooth surface Score=5 Plaque coverage over more than two third of the tooth surface.
Gingival condition | 0 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975)
Gingival condition | 4 weeks
  Gingival Bleeding Index (Ainamo & Bay, 1975)
Probing depth (PD) | 0 weeks
  Distance from the gingival margin to the base of the pocket (mm)
Probing depth (PD) | 4 weeks
  Distance from the gingival margin to the base of the pocket (mm)
Recession (REC) | 0 weeks
  Distance from the gingival margin to the cemento-enamel junction (mm)
Recession (REC) | 4 weeks
  Distance from the gingival margin to the cemento-enamel junction (mm)
Patient-reported outcome measures (PROMs) | 2 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, and also on possible factors influencing tooth staining, such as the consumption of certain foods and drinks, as well as compliance with product use.
Patient-reported outcome measures (PROMs) | 4 weeks
  A predefined questionnaire will be filled by the patient, on product usage and perceptions, and also on possible factors influencing tooth staining, such as the consumption of certain foods and drinks, as well as compliance with product use.
Compliance | 2 weeks
  The study coordinator will collect, at each study visit, the compliance forms, filled by the patients, as well as the empty and unused tubes and mouth rinse bottles. In the compliance forms, information about the number of times a day has the patient used the dentifrices and the rinses during the whole study period will be recorded.
Compliance | 4 weeks
  The study coordinator will collect, at each study visit, the compliance forms, filled by the patients, as well as the empty and unused tubes and mouth rinse bottles. In the compliance forms, information about the number of times a day has the patient used the dentifrices and the rinses during the whole study period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David Herrera, Prof., Principal Investigator — Etiology and Therapy of Periodontal and Periimplant Research Group (ETEP). Faculty of Dentistry. University Complutense of Madrid (UCM)
Locations (1):
- Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No